CLINICAL TRIAL: NCT01421862
Title: The Genetics of "Non-Response" in Adult AML
Brief Title: Biomarkers in Samples From Adult Patients With Acute Myeloid Leukemia Who Failed Existing Standard-of-Care Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Jerry Radich, Fred Hutchinson Cancer Research Center
Other Study IDs: FHCRC-9140; CDR0000709269 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2011-08-20; First posted 2011-08-23 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2011-08

CONDITIONS: Leukemia
Keywords: adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; adult acute myeloblastic leukemia without maturation (M1); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities; Leukemia, Megakaryoblastic, Acute | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Base Sequence

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer who failed treatment may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer resistance. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies biomarkers in samples from adult patients with acute myeloid leukemia who failed standard-of-care treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define a "non-response" signature that will help up-front identification of cases of intermediate-risk acute myeloid leukemia (AML) destined to fail existing standard-of-care therapy.
* Identify biological pathways in the "non-response" group that can provide targets for novel therapeutics.

OUTLINE: DNA and RNA extracted from cryopreserved bone marrow cells and/or blood cells are analyzed for mutations and gene expression signatures (genome-wide methylation, mRNA and miRNA expression, and single nucleotide polymorphism (SNP) analysis) by microarray assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples from previously untreated non-M3 acute myeloid leukemia (AML)
* Normal karyotype (NK) intermediate-risk disease
* Two or more vials of cryopreserved pretreatment bone marrow cells and/or two or more vials of cryopreserved pretreatment blood cells available from the Intergroup AML Repository
* Blast count ≥ 60%
* Eligible and evaluable for the patient's clinical trial, and did not have fatal induction toxicity
* Response to protocol induction chemotherapy:

  * Non-response: AML with failure to achieve a complete remission (CR) after induction chemotherapy ("7 & 3"-based therapy using cytatabine and/or daunorobicin hydrochloride (DNR) OR idarubicin and/or DNR
  * Responders: continued complete remission (CCR) > 2 years

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Genetic signature predictive of progression and drug resistance in AML

SECONDARY OUTCOMES:
Identification of biological pathways in non-responder AML patients

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Radich, MD, Principal Investigator — Fred Hutchinson Cancer Center